CLINICAL TRIAL: NCT00001129
Title: Adherence Strategies Using a Medication Manager and an Electronic Medication Reminder System for HIV-Infected Patients Receiving HAART
Brief Title: A Study of Two Adherence Plans to Help HIV-Positive Patients Take Their Medications Correctly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Model: Factorial | Purpose: Treatment
Other Study IDs: CPCRA 062; 11617 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2000-01-17; First posted 2001-08-31 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; RNA, Viral; Patient Compliance; Anti-HIV Agents; Viral Load; Reminder Systems; Treatment Experienced; Treatment Naive
MeSH Terms: conditions — HIV Infections; Patient Compliance

INTERVENTIONS:
Device: Electronic Medication Reminder System
Behavioral: Medication Manager

SUMMARY:
The purpose of this study is to look at different ways to help patients follow their anti-HIV medication schedules.

It is very important that HIV-positive patients take their anti-HIV medications correctly so they get the best possible benefit from them. Taking the drugs correctly, called "adherence," may keep HIV virus levels in the blood (viral load) low for a longer time. However, anti-HIV medication schedules are often complicated, and many patients have difficulty remembering to take their drugs at the correct time. This study will look at 2 different ways to teach patients about the importance of taking their medications correctly and to remind them when to take their medications.

DETAILED DESCRIPTION:
Adherence to antiretroviral (AR) therapy has become increasingly important in the management of HIV infection. Adherence to AR regimens is thought to be a critical factor in maintaining therapeutic drug levels, thus helping ensure viral suppression and minimizing the risk of drug resistance. However, AR regimens are often complex with demanding dosing schedules. Patients often miss doses because they simply forget; other factors such as substance abuse, depression, and low literacy levels also contribute to nonadherence. Adherence is influenced not only by individual behavior but also by the services, the quality of the patient-provider relationship, and the amount of social support offered the patient. There is no currently agreed upon, widely used, and generalizable intervention for improving adherence over the long course of HIV therapy. This study provides a long-term comparative evaluation of two interventions.

Clinical sites, rather than individual patients, are randomized to one of four groups: a medication manager, an electronic medication reminder system, a medication manager plus an electronic medication reminder system, or usual care. Special training sessions are held for the staff of participating units assigned to medication manager and/or electronic medication reminder system interventions. The medication manager is a research staff member who works individually with study patients, addressing the knowledge, motivation, and skills necessary for adherence. The electronic medication reminder system is ALR (A Little Reminder). This is a small, portable alarm that is programmed to sound and flash at the times of the patient's scheduled AR medication doses. Patients enrolling into either the FIRST or MDR-HIV study at clinical sites authorized to carry out this study are offered the option of participating in the adherence intervention to which the clinical site has been randomly assigned. Data collected through the FIRST and the MDR-HIV protocols are used to address the Adherence study objectives. Patients on the FIRST protocol are assessed for time to first plasma HIV-RNA level above 2,000 copies/ml. Also, patients on the FIRST and MDR-HIV studies are assessed for changes in viral load, resistance, CD4 cell counts, adherence, and other factors.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are enrolling in a qualifying CPCRA AR therapeutic study. Currently, the FIRST and MDR-HIV studies are the only qualifying protocols.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Are enrolling at a clinic site that is unable to participate in this study for some reason.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1248
Dates: Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Mannheimer, Study Chair; Edward Morse, Study Chair
Locations (20):
- United States (20):
  - Community Consortium / UCSF, San Francisco, California
  - Virginia Cafaro M.D., San Francisco, California
  - Denver CPCRA / Denver Public Hlth, Denver, Colorado
  - Univ Hosp Infectious Diseases Clinic, Denver, Colorado
  - Yale Univ School of Medicine / AIDS Program, New Haven, Connecticut
  - Washington Reg AIDS Prog / Dept of Infect Dis, Washington D.C., District of Columbia
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - AIDS Research Alliance - Chicago, Chicago, Illinois
  - Louisiana Comm AIDS Rsch Prog / Tulane Univ Med, New Orleans, Louisiana
  - Wayne State Univ - WSU/DMC / Univ Hlth Ctr, Detroit, Michigan
  - Henry Ford Hosp, Detroit, Michigan
  - Southern New Jersey AIDS Clinical Trials, Camden, New Jersey
  - North Jersey Community Research Initiative, Newark, New Jersey
  - Partners in Research / New Mexico, Albuquerque, New Mexico
  - Harlem AIDS Treatment Grp / Harlem Hosp Ctr, New York, New York
  - Bronx-Lebanon Hosp Ctr, The Bronx, New York
  - The Research and Education Group, Portland, Oregon
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Univ TX Health Science Ctr, Houston, Texas
  - Richmond AIDS Consortium / Div of Infect Diseases, Richmond, Virginia